CLINICAL TRIAL: NCT05285592
Title: Fecal Microbiota Therapy in Steroid Ineligible Alcoholic Hepatitis: A Randomized Controlled Trial.
Brief Title: Fecal Microbiota Therapy in Steroid Ineligible Alcoholic Hepatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Alcoholic Hepatitis-02
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Transplantation (Experimental): 1. Donors will be supplied clean, sealable containers for collection and transport of stool. Containers will be labeled with the name, UHID and date/time of stool collection.
  2. Collected stool will be immediately transferred to the laboratory facility for processing and used within 6 hours collection
  3. Stool sample from Healthy donor will be processed
  4. Patient preparation
  5. Patient was kept NPO for 4 hours prior to stool instillation
  6. Iv antibiotics were continued as per treating doctor in the event of sepsis
  7. The patient was allowed to consume the prescribed diet 2 hours after the procedure instillation
  8. Methods of FMT infusion.
  9. Seven doses (30gm one dose) of FMT will be given via jejunal port of NJ/NG tube
  Interventions: Other: Fecal Transplantation
- Standard Medical Treatment (Active Comparator): Standard Medical Treatment
  Interventions: Drug: Standard Medical Treatment

INTERVENTIONS:
Other: Fecal Transplantation — Fecal Transplantation
  Arms: Fecal Transplantation
Drug: Standard Medical Treatment — Standard Medical Treatment
  Arms: Standard Medical Treatment

SUMMARY:
Alcoholic hepatitis, the most florid form of alcoholic liver disease, has a very high short-term mortality of up to 50% and no specific therapies are available other than steroids. Steroids also only show a limited utility in improving the short-term survival and boast no evidence of any long-term benefits. Additionally, only a small proportion of patients with alcoholic hepatitis are eligible to receive steroids. Thus, a large number of patients are either not eligible or do not respond to steroids and this group outnumbers those who do respond to steroids, leaving us without any specific therapeutic options for a majority of these individuals.Even liver transplantation is not feasible in most cases due to the presence of sepsis or recent alcohol consumption and many ethical and logistic issues are involved despite the documented safety and survival benefits of early liver transplantation in patients with severe alcoholic hepatitis (SAH) not responding to medical management.Therefore, newer, more effective, and nontransplant therapeutic options for managing severe alcoholic hepatitis are needed. Since gut dysbiosis, leaky gut, and products of the gut microbiome reaching the liver are the main culprits in the development of alcoholic hepatitis, targeting qualitative and quantitative changes in the gut microbiome remains an important strategy in developing new therapies for alcoholic hepatitis. Among others, the modulation of gut microbiota by fecal microbiota transplantation (FMT) has recently been conceptualized and evaluated as a potential therapeutic strategy in both preclinical and clinical studies.

DETAILED DESCRIPTION:
AIM- To assess survival benefit at 3 month, in patients of severe alcoholic hepatitis who are steroid ineligible.

Methodology:

Study population: Fecal microbiota therapy in steroid ineligible Alcoholic hepatitis: Randomized controlled trial.

Study design:

A prospective, randomized controlled trial. The study will be conducted on the consecutive patients presenting with severe Alcoholic hepatitis to the wards of Department of Hepatology, ILBS, New Delhi from feb 2022 to February 2023 who meet the inclusion criteria.

Study period: 2 years from the date of ethics approval

Techinue for FMT Healthy donor will be screen as per ILBS FMT proforma- donor should be from family and emotionly attached.

Stool collection

1. Donors will be supplied clean, sealable containers for collection and transport of stool. Containers will be labeled with the name, UHID and date/time of stool collection.
2. Collected stool will be immediately transferred to the laboratory facility for processing and used within 6 hours collection
3. Stool sample from Healthy donor will be processed
4. Patient preparation
5. Patient was kept NPO for 4 hours prior to stool instillation
6. Iv antibiotics were continued as per treating doctor in the event of sepsis
7. The patient was allowed to consume the prescribed diet 2 hours after the procedure instillation
8. Methods of FMT infusion.
9. Seven doses (30gm one dose) of FMT will be given via jejunal port of NJ/NG tube

Sample size with justification:

Assuming that the survival in FMT group is 87.5% and 33% in SMT Group with alpha 5 %, power 95% we need to enroll 52 in FMT group and 26 in SMT Group so that the FMT versus SMT ration is 2. Further assuming 5% defaulter rate /drop out rate we decided to enroll 56 and 28 on FMT and SMT arm.We will enroll 84 patients, block size of 6

Intervention:

1. Patients will be randomized into two Arms A & B.
2. Arm A will receive fecal microbioata therapy for 7 Days, Seven doses (30gm stool prepared in 100 ml Ns everyday as described ) of FMT will be given via jejunal port of NJ/NG tube.
3. Arm B will receive standard medical therapy.
4. Patient preparation in Arm A
5. Patient was kept NPO for 4 hours prior to stool instillation
6. Iv antibiotics were continued as per treating doctor in the event of sepsis
7. The patient will be allowed to consume the prescribed diet 2 hours after the procedure.
8. Both groups received Antibiotics, multivitamins, albumin infusions, nutrition will be used as per clinical discretion in both groups.

Data to be collected:

1. Baseline - CBC, LFT, RFT, Serum albumin, total protein, Chest X Ray, Serum electrolytes, PT, INR baseline and then for first 7 days then at 28 days ,90 and 180 days then whenever needed
2. PCT and CRP baseline and whenever needed
3. Amylase, lipase baseline if needed
4. HIV,IgM,HAV Ab,IgM HEV, HBsAg, HB core Ab (total),AntiHCV- baseline
5. Blood cultures x2- baseline and whenever needed
6. Urine culture & urinalysis-Baseline and whenever needed
7. Ascites for albumin, total protein, TLC cell count and differential, SAAG, G/S, C/s (if present)
8. TNF alpha, TGF B, IL 1, IL 6, IL22 baseline then at 28 days,90 and 180 days.
9. Stool studies (if diarrhea): C. difficile, culture,
10. stool Microbioata analysis baseline and whenever needed
11. Glucose H2 Breath test if needed
12. UGI endoscopy with (D2 biopsy/Aspirate whenever feasible), and NJ placement done at baeline for FMT insertion.
13. Complete abdominal ultrasound or cross-sectional radiology
14. Liver Biopsy (If Feasible)

Statistical Analysis:

Data will be reported as mean + SD. Categorical variables will be compared using the chi-square test or Fisher exact test. Normal continuous variables will be compared using the Student's t test Non normal continuous variables will be compared using the Mann Whitney rank-sum test (unpaired data) or the Wilcoxon test (paired data). The actuarial probability of survival will be calculated by the Kaplan-Meier method and compared using the log-rank test. A Cox regression analysis will be performed to identify independent prognostic factors for survival.Univariate and multivariate analysis will be used whenever applicable.

Adverse effects:

Side effects related to FMT will be noted. Abdominal Pain, Bloating, loss of appetite Gas/Flatulence, Constipation, Diarrhea , Nausea ,Vomiting Fever

Stopping rule of study:

1. New onset infection (sepsis)
2. Patient refusal After starting Therapy
3. Liver transplantation

Expected outcome of the project-Modulation of gut microbiota and correction of dysbiosis in severe Alcoholic hepatitis through healthy donor Fecal Implantation therapy improves gut dysbiosis and provide survival benefit at 3 months

ELIGIBILITY:
Inclusion Criteria:

1. Steroid ineligible severe alcoholic hepatitis as per definition
2. Informed consent
3. Age 18 - 70 years
4. Liver biopsy -if Feasible
5. Model for End-Stage Liver Disease (MELD) ≥ 20 and Maddrey DF ≥ 32

Exclusion Criteria:

1. UGI Bleed within last one month
2. More then 3 organ failure requiring support
3. Mechanically ventilated patient , (patients requiring ICU/ HDU care) (On inotropic support)
4. Uncontrolled sepsis, DIC
5. Gut paralysis
6. Active hepatic or extra hepatic malignancy
7. Renal failure creatinine > 2.5
8. DF>120
9. MELD >35
10. Prior SBP/active SBP
11. Intestinal conditions like IBD, SIBO

Donor evaluation The subjects will be screened for

1. Routine laboratory tests (CBC; LFT; KFT; PT; INR)
2. Fasting blood sugar
3. Lipid profile
4. HBsAg
5. Anti-HCV
6. HIV 1 & 2
7. VDRL
8. Stool routine and microscopy stool ova & cysts.
9. Stool culture
10. Clostridium difficile toxin
11. Helicobacter pylori stool antigen
12. Cryptosporidium & Isospora (acid fast stain) Exclusion criteria for Donor

1. Antibiotic usage within 3 months of enrollment 2. Gastroenteritis within last 2 months 3. Obesity 4. Diabetes mellitus 5. Inflammatory bowel disease 6. Any Malignancy 7. Chronic Kidney disease, Coronary artery disease 8. Cerebrovascular accident or chronic obstructive pulmonary disease 9. HBsAg, Anti HCV, HIV seropositivity 10. Transaminitis, dyslipidemia 11. Ova or cyst in stool, C. difficile toxin Positive 12. Chronic alcohol intake 13. Active substance abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Mortality at 3 months | 3 months
Liver transplant free survival | 3 months

SECONDARY OUTCOMES:
End of study period | 6 months
Mortality | 1 month
Post therapy assessment in the form of clinical improvement (hepatic encephalopathy, ascites , improvement in jaundice)(both ascites and HE if present) | 6 months
Frequency of decompensation events on follow up period | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided